CLINICAL TRIAL: NCT00427947
Title: Continuous Popliteal Sciatic Nerve Block Interest in Postoperative Pain Management for Patients With Leg Amputation
Brief Title: Leg Amputation and Continuous Sciatic Nerve Block
Acronym: CAPDAF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of patients
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9440-05; 2004-037
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Phantom Limb; Leg Amputation
Keywords: phantom limb pain; amputation; anesthetics, local; postoperative analgesia; ropivacaine; analgesia
MeSH Terms: conditions — Phantom Limb; Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Continuous sciatic nerve bloc : ropivacaine infusion
  Interventions: Drug: ropivacaine/placebo
- 2 (Placebo Comparator): Continuous sciatic nerve bloc : NaCl Infusion
  Interventions: Drug: ropivacaine/placebo

INTERVENTIONS:
Drug: ropivacaine/placebo — Continuous sciatic nerve bloc

SUMMARY:
Analgesia following leg amputation is based on morphine administration. For elderly patients of ASA physical status 2 or 3, morphine sparing is possible when perinervous block techniques are used. Phantom limb pain complicates leg amputation in 50 to 80% of cases. Prevention of these pains has been studied in various clinical trials but the interest of perinervous block technique remains to be evaluated.

The purpose of the study is to evaluate the benefit of perioperative locoregional analgesia by ropivacaine via a popliteal sciatic catheter on intravenous morphine consumption during the 72 first postoperative hours following leg (below knee) amputation The study will be randomized, double blinded, controlled clinical trial and 84 patients undergoing leg amputation (below knee) will be included Patients will be divided into 2 groups: one group of patients who will benefit perioperative locoregional analgesia by ropivacaine via a popliteal sciatic catheter and morphine for analgesia and the other one who will benefit placebo through the catheter and morphine.

The investigators will evaluate the efficacy of the continuous popliteal sciatic nerve block in postoperative analgesia after leg amputation and prove the efficacy of a perioperative analgesia by continuous popliteal sciatic nerve block to prevent phantom limb pain after leg amputation in patients of ASA physical status 2 or 3.

DETAILED DESCRIPTION:
Introduction:

Analgesia following leg amputation is based on morphine administration. For elderly patients of ASA physical status 2 or 3, morphine sparing is possible when perinervous block techniques are used. Indeed, per operative placement of a perinervous catheter by the surgeon allows a morphine consumption decrease of about 30%. Nevertheless, the interest of a sciatic block providing analgesia in the tibial and fibular territories has still to be assessed in this indication.

Phantom limb pain complicates leg amputation in 50 to 80% of cases. Risk factors of this complication are numerous, from central or peripheral origin. Phantom limb pain postpones patients' social and professional rehabilitation, and results in an increased medical consumption. Prevention of these pains has been studied in various clinical trials, and results need confirmation. Thus, epidural analgesia alone does not decrease the long term incidence of phantom limb pain.

Objectives:

Primary : To compare intravenous morphine consumption during the 72 first postoperative hours following leg (below knee) amputation of patients randomly assigned in two groups. One group benefit from perioperative locoregional analgesia by ropivacaine via a popliteal sciatic catheter, the other group is given placebo through the catheter.

Secondary :

* To assess tolerance and adverse effects (myalgia, infection, adverse effects of local anaesthetics) of the popliteal sciatic catheter during the 72 first postoperative hours and on the 7th postoperative day, in patients with ASA physical status 2 or 3
* To compare tolerance and adverse effects of morphine during the protocol in the 2 groups of patients
* To assess the long term effects of the preoperative continuous popliteal sciatic nerve block: incidence of stump pain and phantom limb pain, time of outbreak, intensity (VAS), characteristics (French version of the McGill Pain Questionnaire and DN4 questionnaire), and the analgesic consumption over a year.
* To assess the possibility for the patients to use a prosthesis

Population:

Eighty four patients scheduled for leg amputation (below knee), randomly allocated in 2 groups of forty patients, according to the type of analgesia. Patients were enrolled in the general and vascular surgery unit, CHU (University Hospital) Pellegrin Bordeaux.

Methods:

Randomised clinical trial, with two parallel groups, with direct individual benefit, double-blinded, realised on a population of patients undergoing leg amputation, comparing different clinical parameters of postoperative pain evaluation, and outbreak of phantom limb pain according to the group of analgesia.

* One group of patients with locoregional analgesia associated with morphine administration (assessed treatment)
* One group of patients with morphine analgesia only (reference treatment). Patients will be followed for one year. This study will last 3 years in a general and vascular surgery unit, inclusion will be realised during 34 months by anaesthetists and surgeons, an extension of this study for one year will be done with the objective of a cohort follow-up.

Statistical analysis will be done with intention to treat.

Anticipated results:

To prove the efficacy of the continuous popliteal sciatic nerve block in postoperative analgesia after leg amputation.

To prove the efficacy of a perioperative analgesia by continuous popliteal sciatic nerve block to prevent phantom limb pain after leg amputation in patients of ASA physical status 2 or 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for leg amputation following arteritis
* ASA score: 2-3
* Informed consent obtained from the patient

Exclusion Criteria:

* Patients involved in another clinical trial
* Post-infection OR post traumatic leg amputation
* Blood coagulation disorders
* Local anesthetic, morphine, or paracetamol allergy
* Local inflammatory signs
* Pregnant or breastfeeding women
* Patients with protective supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-12; Primary Completion 2009-04 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Total intravenous morphine consumption | during the first 72 postoperative hours following leg (below knee) amputation

SECONDARY OUTCOMES:
tolerance and adverse effects (myalgia, infection, adverse effects of local anaesthetics) of the popliteal sciatic catheter, in patients with ASA physical status 2 or 3 | during the 72 first postoperative hours and on the 7th postoperative day
tolerance and adverse effects of morphine during the protocol in the 2 groups of patients | during the first 72 postoperative hours
incidence of stump pain and phantom limb pain, time of outbreak, intensity (VAS), characteristics (French version of the McGill Pain Questionnaire and DN4 qu | 1, 3, 6 and 12 months postoperative
use of prosthesis | 1, 3, 6 and 12 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Karine NOUETTE GAULAIN, Dr, Principal Investigator — University Hospital, Bordeaux, France; Antoine BENARD, Dr, Study Chair — university hospital, Bordeaux, France
Locations (1):
- Département d'anesthésie réanimation I, Hopital Pellegrin, CHU de Bordeaux, Bordeaux, France